CLINICAL TRIAL: NCT01731522
Title: Eating Frequency Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Tennessee, Knoxville (Other)
Responsible Party: Principal Investigator, Hollie Raynor, Professor, The University of Tennessee, Knoxville
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: MTRI-Basic EF Study
Record Dates: First submitted 2012-11-14; First posted 2012-11-21 (Estimated); Last update posted 2025-04-03 (Actual); Status verified 2025-04

CONDITIONS: Eating Frequency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- EF condition (Experimental)
  Interventions: Behavioral: EF condition

INTERVENTIONS:
Behavioral: EF condition
  Other Names: Grazing, Three meal

SUMMARY:
The purpose of this study is to examine the influence of two Eating Frequency prescriptions, meal (energy intake occurring during three meals per day) and grazing (energy intake occurring every two to three hours per day), on consumption during an ad libitum meal consumed at the end of the day, overall daily energy intake, and ratio of energy intake to energy expenditure. It is hypothesized that the grazing condition will produce lower consumption during an evening ad libitum meal, lower daily energy intake, and a lower ratio of energy intake to energy expenditure than the meal condition.

DETAILED DESCRIPTION:
20 men and women of healthy weight will participate in this study. The complete study design will be a 2 x 2 mixed factorial design, with the between-subject factor of order and a within-subject factor of eating condition (meal or grazing). Depending upon the eating condition, participants will be provided with a morning meal and an afternoon meal (meal) or two small meals and three snacks to be consumed every 2-3 hours (grazing). The types of foods and amount of foods provided to participants will be identical in each condition; the only difference in the conditions is the time spacing during the day when the foods are consumed. The primary dependent variable will be amount, both grams and energy, of food consumed during an ad libitum meal consumed in the evening at the completion of the meal condition, overall daily energy intake, and ratio of daily energy intake to energy expenditure. It is hypothesized that the grazing condition will produce lower consumption during an evening ad libitum meal, lower daily energy intake, and a lower ratio of energy intake to energy expenditure than the meal condition.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 35 years
* body mass index (BMI) between 18.5 and 24.9 kg/m2
* no history of overweight or obesity
* unrestrained eater (<12 on Three Factor Eating Questionnaire [TFEQ])
* regularly participate in at least 150 minutes of moderate-intense physical activity per week over the previous 4 weeks

Exclusion Criteria:

* currently taking medication that affects appetite or food intake
* have a medical condition affecting eating or currently following a therapeutic diet
* are currently participating in a weight loss program and/or taking weight loss medication
* have gained or lost > 5% of body weight during the past 6 months
* diagnosed with type 1 or 2 diabetes
* have had bariatric surgery
* report disliking foods used in the investigation (scoring a 1 or 2 on a 5-point Likert scale)
* report having allergies to foods used in the investigation
* currently smoke
* report binge eating
* are graduate students in the Department of Nutrition
* are pregnant, lactating, < 6 months post-partum.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2012-12 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Total grams of ad libitum meal consumed | 1 year
  The foods that will be used in this investigation are Tyson Chicken Breast Tenders, Ore-Ida Tater Tots, Birds Eye Steamfresh Pure & Simple green beans, and Sarah Lee Butter Pound Cake. Participants will be provided with ad libitum amounts of the foods, and the foods will be measured in grams to the tenth decimal point on an electronic food scale (Denver Instrument Co., Arvada, CO) before and after the meal. The weight of the container will also be measured. Total grams of each food consumed during the session will be determined by subtracting pre- and post-consumption weight of food.

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Tennessee-Knoxville, Knoxville, Tennessee, United States